CLINICAL TRIAL: NCT05723874
Title: The Effect of Multiple Oral Doses of Bosentan on the Steady State Kinetics of BI 425809 After Oral Administration to Healthy Male Subjects (an Open-label, Two-period Fixed Sequence Trial)
Brief Title: A Study in Healthy Men to Test Whether Bosentan Influences the Amount of BI 425809 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1346-0056; 2021-006676-17 (EudraCT Number)
Record Dates: First submitted 2023-01-31; First posted 2023-02-13 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-10

CONDITIONS: Healthy
MeSH Terms: interventions — BI 425809; Bosentan

STUDY DESIGN:
Intervention Model Description: Patients cross over from reference treatment (R) to test treatment (T) (two periods, fixed sequence).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BI 425809 (reference treatment, R) then BI 425809 + bosentan (test treatment, T) (Experimental)
  Interventions: Drug: BI 425809; Drug: Bosentan

INTERVENTIONS:
Drug: BI 425809 — BI 425809
  Other Names: Iclepertin
Drug: Bosentan — Bosentan
  Other Names: Tracleer®

SUMMARY:
The main objective of this trial is to investigate the relative bioavailability of BI 425809 given alone (Reference) compared to a combined administration with the moderate CYP3A4 inducer bosentan (Test) following repeated oral administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Age of 30 to 55 years (inclusive)
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive)
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial

Exclusion Criteria:

* Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
* Repeated measurement of systolic blood pressure outside the range of 90 to 140 mmHg, diastolic blood pressure outside the range of 50 to 90 millimetre of mercury (mmHg), or pulse rate outside the range of 45 to 90 beats per minute (bpm)
* Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
* Any evidence of a concomitant disease assessed as clinically relevant by the investigator
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
* History of relevant orthostatic hypotension, fainting spells, or blackouts
* Further exclusion criteria apply

Ages: 30 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-05-26 (Actual); Study Completion 2023-05-26 (Actual)

PRIMARY OUTCOMES:
Area under the concentration-time curve of the analyte in plasma at steady state over a uniform dosing interval τ (AUCτ,ss) | On Day 10 of period 1 and on Day 14 of period 2.
Maximum measured concentration of the analyte in plasma at steady state over a uniform dosing interval τ (Cmax,ss) | On Day 10 of period 1 and on Day 14 of period 2.

SECONDARY OUTCOMES:
Minimum concentration of the analyte in plasma at steady state within a uniform dosing interval τ (Cmin,ss) | On Day 10 of period 1 and on Day 14 of period 2.

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com